CLINICAL TRIAL: NCT00351091
Title: a Six Month, Multicenter, Randomized, Double-blind, Active-controlled, Parallel Group Study to Estimate the Pharmacodynamic Response of Two Risedronate Regimens Compared With 5mg Daily : 150mg Monthly Dose for Six Months and 15mg Daily for Thirty Days Followed by 150mg Monthly Dose for 5 Months in Postmenopausal Women With Low Bone Density.
Brief Title: Risedronate in Postmenopausal Women With Low Bone Density
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMR4003B_2501
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: OSTEOPOROSIS, POSTMENOPAUSAL
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: RISEDRONATE

SUMMARY:
The primary objective of this pilot study is to estimate the percent change from baseline at Week 4, Month 6 in NTX bone turnover marker for a monthly 150mg dose of risedronate administered for 6 months and a loading dose regimen of risedronate over a 6 month treatment period both compared to a 5 mg daily dose of risedronate for 6 months

The secondary objectives are :

* To estimate the percent change from baseline at specified visits other than Week 4, Month 6 in NTX for the monthly 150 mg dose of risedronate administered for 6 months and the loading dose regimen of risedronate over a 6 month treatment period both compared to the 5 mg daily dose of risedronate.
* To estimate the percent change from baseline at all specified visits in serum CTX and bone specific alkaline phosphatase for the monthly 150 mg dose of risedronate administered for 6 months and the loading dose regimen of risedronate over a 6 month treatment period both compared to the 5 mg daily of risedronate.
* To estimate the percent change from baseline at Month 6 in lumbar spine BMD for the monthly 150 mg dose of risedronate administered for 6 months and the loading dose regimen of risedronate over a 6 month treatment period both compared to the 5 mg daily dose of risedronate.
* To evaluate the safety of the risedronate 150 mg monthly and the loading dose regimen.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory women,postmenopausal >= 5 years
* have lumbar spine baseline BMD within the following criterion :

  * Hologic: <= 0.827 g/cm2 or
  * Lunar: <= 0.942 g/cm2 or
  * Norland: <= 0.768 g/cm2
* be in general good health as determined by medical history, physical examination and laboratory tests

Exclusion Criteria:

* serum 25-OH vitamin D level <= 12 ng/ml
* history of osteomalacia
* history of active hyperparathyroidism or hyperthyroidism
* hypocalcemia or hypercalcemia from any cause
* depot injection >10,000 IU Vitamin D in the past 9 months prior to starting the investigational product
* use of Vitamin D supplementation within 3 months prior to starting the investigational product
* use of any of the following medications within a specified number of months prior to starting the investigational product :

  * any bisphosphonate.
  * use of any fluoride with the exception of fluoride use for oral hygiene
  * strontium
  * other bone active agents
  * subcutaneous estrogen implant
  * oral or parenteral glucocorticoids
  * anabolic steroids
  * estrogen or estrogen-related drugs, except for low dose vaginal creams
  * progestogen
  * calcitonin, calcitriol, or calcifediol
* any allergic or abnormal reaction to bisphosphonates
* creatinine clearance < 30 ml/min

Ages: 65 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2002-11; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Urine NTX at week 4 of month 6

SECONDARY OUTCOMES:
Urine NTX at other visits, serum CTX and bone specific alkaline phosphatase, lumbar spine BMD

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi